CLINICAL TRIAL: NCT03317275
Title: Diagnostic Value of 18F-Fluoride-PET/MRI in the Management of Suspected Facet Joint Arthropathy: A Prospective Cohort Study
Brief Title: Diagnostic Value of 18F-Fluoride-PET/MRI in the Management of Suspected Facet Joint Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PET/MRI
Record Dates: First submitted 2017-06-07; First posted 2017-10-23 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Arthropathy of Lumbar Facet; Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomised cohort study, partial blinded
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection based on 18F-Fluoride-PET/MRI (Experimental): One group will undergo facet injection(s) according to the 18F-Fluoride-PET/MRI result, with standard injections performed under CT-guidance. The Pain assessment by VAS immediately before the facet joint injection, at 15 minutes, 1 day, 1 week and 1 month after the injection, as performed routinely in our institution.
  Interventions: Device: 18F-Fluoride-PET/MRI; Procedure: facet injection; Other: pain assessment by VAS
- injection based on clinical practise (Active Comparator): The control group will undergo facet injections blinded to the 18F-Fluoride-PET/MRI results, but based on current standard clinical practise (MRI and clinical correlation). Pain assessment by VAS immediately before the facet joint injection, at 15 minutes, 1 day, 1 week and 1 month after the injection, as performed routinely in our institution.
  Interventions: Device: 18F-Fluoride-PET/MRI; Procedure: facet injection; Other: pain assessment by VAS

INTERVENTIONS:
Device: 18F-Fluoride-PET/MRI — facet joint injection guided by the anatomical localization of causative structures by PET/MRI compared to standard assessment techniques.
Procedure: facet injection — facet joint local anesthetic and corticosteroid injection according to the 18F-Fluoride-PET/MRI result or based on current standard clinical practise (MRI and clinical correlation) respectively
Other: pain assessment by VAS — VAS questionnaire immediately before the facet joint injection, at 15 minutes, 1 day, 1 week and 1 month after the injection, as performed routinely in our institution.

SUMMARY:
Prior to the injection, the facet joints have to be defined according to standard radiological techniques (e.g. MRI and physical correlation). Patients are then sent to 18F-Fluoride-PET/MRI imaging, in order to localize facet joints with increased uptake. Facet joints to be injected are again defined according to the location(s) of highest uptake as demonstrated by 18F-Fluoride-PET/MRI.

The defined injection sites before and after PET/MRI are compared. In equal defined injection sites, patients are sent for infiltration as scheduled, otherwise patients are randomized into two groups.

One group will undergo facet injection(s) according to the 18F-Fluoride-PET/MRI result, with standard injections performed under CT-guidance by the radiology department of the study site. The control group will undergo facet injections blinded to the 18F-Fluoride-PET/MRI results, but based on current standard clinical practise (MRI and clinical correlation).

The patients are asked to complete a validated pain and function questionnaire immediately before the facet joint injection, at 15 minutes, 1 day, 1 week and 1 month after the injection, as performed routinely in our institution.

The purpose of this study is to prospectively evaluate the value of 18F-Fluoride-PET/MRI imaging in patients with low back pain with evidence of painful facet joint arthropathy, which would potentially benefit from facet joint injections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old with low back pain who have failed conservative management in the primary care setting, namely, analgesia and physical therapy.
2. Imaging evidence (e.g. MRI) of facet joint degeneration, such as facet hypertrophy, subchondral sclerosis, and joint space narrowing.
3. Obtained informed consent

Exclusion Criteria:

1. had undergone prior spinal surgery or prior facet joint injections or
2. had other spinal abnormalities (benign or malignant tumors, congenital defects, isthmic spondylolisthesis) or
3. are unable to tolerate PET/MRI imaging
4. are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
pain reduction | VAS immediately before the facet joint injection, at 15 minutes, 1 day, 1 week and 1 month after the injection
  reduction of pain after facet joint injection assessed by visual analogue scale (VAS)

SECONDARY OUTCOMES:
location of uptake in 18F-Fluoride-PET/MRI | 40 +/- 7 days post injection
  location of uptake in 18F-Fluoride-PET/MRI assessed by radiologist
quantity of uptake in 18F-Fluoride-PET/MRI | 40 +/- 7 days post injection
  quantity of uptake in 18F-Fluoride-PET/MRI assessed by radiologist

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, PD Dr. med., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Clinic Balgrist, Zurich, Canton of Zurich, Switzerland